CLINICAL TRIAL: NCT06498986
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 in Combination With Osimertinib Mesylate Tablets in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of BL-B01D1 in Combination With Osimertinib Mesylate Tablets in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-207
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1+Osimertinib Mesylate Tablets (Experimental): Participants receive BL-B01D1+Osimertinib Mesylate Tablets in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: Osimertinib Mesylate Tablets — Oral administration, 80mg daily for a cycle of 3 weeks.

SUMMARY:
This phase II clinical study is a study to explore the efficacy and safety of BL-B01D1 in combination with Osimertinib Mesylate Tablets in patients with histologically and/or cytologically confirmed locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age ≥18 years old;
4. Expected survival time ≥3 months;
5. Patients with histologically and/or cytologically confirmed locally advanced or metastatic non-small cell lung cancer;
6. Documentation of EGFR sensitive mutations detected from tumor tissue or blood samples;
7. Consent to provide archived tumor tissue or fresh tissue samples from primary or metastatic sites within 2 years for biomarker testing;
8. At least one measurable lesion meeting the RECIST v1.1 definition was required;
9. ECOG ≤1;
10. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
12. The level of organ function must meet the requirements on the premise that blood transfusion is not allowed within 14 days before the screening period and no cell growth factor drugs are allowed;
13. Blood coagulation function: international standardization ratio of 1.5 or less, and the part activated clotting time live enzymes acuities were 1.5 x ULN;
14. Urine protein ≤2+ or ≤1000mg/24h;
15. Fertile female subjects or male subjects with fertile partners must use highly effective contraception from 7 days before the first dose until 6 months after the dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Patients with prior systemic therapy;
2. Previous treatment with EGFR-TKI;
3. Participants who participated in any other clinical trial within 4 weeks before the trial dose;
4. Traditional Chinese medicine (TCM) which had received radiotherapy within 4 weeks before the first use of the study drug and had anti-tumor indications within 2 weeks before the first use of the study drug;
5. Had undergone major surgery within 4 weeks before the first dose;
6. History of severe heart disease or cerebrovascular disease;
7. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
8. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
9. Previous history of interstitial lung disease requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis;
10. Complicated pulmonary diseases leading to clinically severe respiratory function impairment;
11. Severe systemic infection within 4 weeks before screening;
12. Patients at risk for active autoimmune disease or with a history of autoimmune disease;
13. Other malignant tumors within 5 years before the first dose;
14. HIV antibody positive, active tuberculosis, active hepatitis B virus infection, or hepatitis C virus infection;
15. Hypertension poorly controlled by two antihypertensive drugs;
16. Patients with poor glycemic control;
17. Patients with massive effusions, or effusions with obvious symptoms, or poorly controlled effusions;
18. Patients with active central nervous system metastases;
19. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
20. Severe unhealed wound, ulcer, or fracture within 4 weeks before consent signing;
21. Sign a four weeks before there were clinically significant bleeding or bleeding tendency obviously subjects;
22. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
23. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
24. A history of severe neurological or psychiatric illness;
25. Pregnant or lactating women;
26. Subjects who were scheduled to receive live vaccine or received live vaccine within 28 days before study randomization;
27. Other conditions for participation in the trial were not considered appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China